CLINICAL TRIAL: NCT03380715
Title: A Comparison Between Co-phenylcaine Nasal Spray and Nasal Nebulization Prior to Rigid Nasoendoscopic Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: julius
Record Dates: First submitted 2017-11-01; First posted 2017-12-21 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2017-12

CONDITIONS: Anaesthesia; Rhinitis
Keywords: Sinusitis; Endoscopy; Rhinitis
MeSH Terms: conditions — Rhinitis; Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- right nostril in patients with rhinitis (Active Comparator): Intervention : Administration of either 4 sprays of nasal decongestions(Co-Phenylcaine(400mcl) (20mg lidocaine + 2mg phenylephrine) once into the right nasal cavity or
  Interventions: Device: Nasal nebulisation into the right nostril; Device: Nasal Spray into the right nostril
- Left nostril in patients with rhinitis (No Intervention): No nasal decongestion administration into the left nostril
- Right nostril in patients with rhinitis (Active Comparator): 400mcl of co-phenylcaine (20mg of lidocaine + 2mg of phenylephrine) is added into the nasal nebuliser device (Rinowash Nebula, Air liquid medical systems) and the solution is diluted with 4.5cc of isotonic normal saline. This Mixture is then nebulised into the right nasal cavity for approximately 3 minutes.The seated patient's head is kept flexed and nebulizer device is kept sealed within the nasal cavity while the nebulisation is done and subsequently checking nasal resistance after nasal nebulisation.
  Interventions: Device: Nasal nebulisation into the right nostril; Device: Nasal Spray into the right nostril

INTERVENTIONS:
Device: Nasal nebulisation into the right nostril — 400mcl of co-phenylcaine (20mg of lidocaine + 2mg of phenylephrine) is added into the nasal nebuliser device (Rinowash Nebula, Air liquid medical systems) and the solution is diluted with 4.5cc of isotonic normal saline. This Mixture is then nebulised into the right nasal cavity for approximately 3 minutes.The seated patient's head is kept flexed and nebulizer device is kept sealed within the nasal cavity while the nebulisation is done and subsequently checking nasal resistance after nasal nebulisation.
  Arms: Right nostril in patients with rhinitis; right nostril in patients with rhinitis
Device: Nasal Spray into the right nostril — Intervention : Administration of 4 sprays of nasal decongestions(Co-Phenylcaine(400mcl) (20mg lidocaine + 2mg phenylephrine) once into the right nasal cavity using a nasal spray and subsequently checking nasal resistance post nasal spray
  Arms: Right nostril in patients with rhinitis; right nostril in patients with rhinitis

SUMMARY:
Co-phenylcaine is a widely available nasal spray commonly used by otorhinolaryngologists for the purpose of decongestion and local anesthetic prior to a nasoendoscopic or nasopharyngolaryngoscopy. It is often used in the outpatient setting and is also useful for minor procedures. It is unique in its properties because it provides both local anesthetic and decongestive effects on the nasal mucosa hence leading to better visualization of the nasal cavity and better comfort for the patient during the procedure.

Pharmacologically, Co-phenylcaine Forte comprises of a combination of Lignocaine 5% (50mg/ml) and phenylephrine 0.5% (5mg/ml) and is commonly marketed in a 50ml bottle attached to a disposable positive displacement atomizer which avoids contamination by preventing contamination of the nozzle tip by secretions from other patients which are commonly seen in older venturi devices.Its decongestive agent (phenylephrine) acts by influencing the sympathetic vasculature tone via alpha adrenoceptors since its properties are sympathomimetic and oppose vasodilation.As for the local anesthethic component (Lignocaine) , it is an amide local anesthetic which blocks fast voltage gated sodium channels in the cell membrane thus leading to a decrease in sensation when performing a nasoendoscopy. Despite of its advantages, there are also disadvantages in the usage of such a device such as the need for regular change of the nozzle head due to the risk of infection and the high cost of using this device in the long run.

Several studies has demonstrated promising results for the efficacy of nebulized medication and its distribution of medication into the nasal cavity and paranasal sinuses in both healthy individuals and cadaver models.Its advantages over the classical nasal spray include better distribution of medication throughout the nasal cavity and better hygiene due to the ability to change and sterilize the nasal nozzle tip before re-usage.

Very little information is available about the delivery of topical decongestants via nasal nebulization on the pre-endoscopic examination of the nasal cavity. This study aims to compare the efficacy of topical decongestants delivered into the nasal cavity using nasal nebulization against the delivery of topical decongestants using conventional nasal sprays.

DETAILED DESCRIPTION:
Objectives General objectives

• To compare the efficacy of co-phenylcaine (Lignocaine + phenylephrine) in the decongestion and anesthesia of the nasal cavity prior to endoscopic examination using nasal nebulization as the delivery device in comparison to conventional nasal spray.

Specific Objectives

* To objectively assess the degree of nasal patency and nasal inspiratory flow by performing anterior rhinomanometry at pre-procedure and post-procedure at 5, 10, 15, and 30 minutes' interval.
* To objectively assess the blood pressure (BP) and pulse rate (PR) changes throughout the post procedural intervals.
* To subjectively assess the pain scores using the Visual analogue scale (VAS) at pre-procedure and post procedure at 5, 10, 15 and 30 minutes' intervals.
* To subjectively assess the after-taste commonly felt by the patient after the procedure.
* To subjectively assess the patient's NOSE (Nasal Obstruction symptom evaluation) score prior to the commencement of the medication.

Methodology This will be a multicenter, non blinded, prospective, randomized controlled trial on the comparison of delivery of nasal decongestive agent (Co-phenylcaine) into the nasal cavity using nasal sprays and nasal nebulization techniques.

Patients matching the inclusion criteria, when visiting the Otorhinolaryngology clinic of Hospital Tengku Ampuan Rahimah Klang and University Malaya Medical centre (UMMC) who require nasoendoscopy, will be invited to take part in this prospective study over 6 months. An informed consent will be taken detailing the procedure, study conducted and risks involved while participating in the study.

Upon agreeing to participate, the participant's baseline parameters will be recorded.

The baseline parameters will be as follows:

1. Baseline BP ,Age, Gender, Race
2. Baseline BMI/Weight/Height
3. Pre procedure anterior Rhinomanometry reading for NIF (Nasal inspiratory flow), Flow Sum, Flow INC

   1. Anterior rhinomanometer (ATMOS Rhino 31 model, ATMOS Medzintecknik GmbH & Co.KG) is used to document serial changes in nasal air flow throughout the procedure.
   2. Procedure is done with the patient seated,secretions from the nose is cleared prior to the procedure.
   3. Nose adapter and hose for pressure measurement is placed in the opposite nostril.
   4. Mask is pressed on to the face to measure the flow while ensuring good fitting.
   5. The patient is asked to breathe in and out while keeping the mouth closed. The average of 3 readings are documented.

   <!-- -->

   1. Procedure is repeated in the opposite nostril.

2. Baseline NOSE (Nasal obstruction symptom evaluation) score prior to procedure. [Figure 1] 3. VAS (Visual analogue scale) for pain. [Figure2].

1. Painful sensation was induced in the right nasal cavity by probing the mucosa overlying the inferior turbinate 1cm from the anterior end with the ring ended Jobson-Horne Probe.
2. Pressure is maintained for about 1 second and the subject is asked to rate the pain based on the visual analogue scale (VAS).
3. 0 represents "no pain "and 10 represents the "worst pain imaginable".
4. Cut off points for pain VAS recommended are: no pain (0-4mm),mild pain (5-44mm),moderate pain (45-74mm), 75-100mm(severe pain).14

The patient is given a randomized labelled card and is grouped according to the procedure. Group A - Nasal spray, Group B - Nasal nebulizer.

Group A - 4 sprays (400mcl) (20mg lidocaine + 2mg phenylephrine)) of co-phenylcaine are given into the right nostril while keeping the left nostril as a control.

Group B - 400mcl of co-phenylcaine (20mg of lidocaine + 2mg of phenylephrine) is added into the nasal nebulizer device (Rinowash Nebula, Air liquid medical systems) and the solution is diluted with 4.5cc of isotonic normal saline. This Mixture is then nebulized into the right nasal cavity for approximately 3 minutes.The seated patient's head is kept flexed and nebulizer device is kept sealed within the nasal cavity while the nebulization is done.

Post procedure, parameters are recorded 5 minutes, 10 minutes, 15 minutes and 30 minutes post procedure

1. Rhinomanometry readings of both nostrils (Right -tested , Left - Control)
2. Pain VAS score 30 minutes' post procedure.
3. BP and PR repeated at 5,10,15 and 30 minutes' post procedure
4. Rigid Endoscopic examination and VAS based on degree of decongestion and ease of endoscopic passage

Ethical considerations The researchers will seek approval from the National Medical Research and Ethics committee (MREC) of the Ministry of health(MOH), Malaysia via the National Medical Research Registry (NMRR). All responses are confidential; all respondents are allowed to refuse participation in the study.

Since both medical devices delivers the same drug,the side effects which the participant may experience include tremors, palpitations, nausea, vomiting, dizziness, numbness and most commonly a transient bitter taste in the mouth for a few minutes. Rarely, the participant may develop a hypersensitive reaction towards the offending medication.The risks will be managed accordingly and symptomatically and the medication will be stopped immediately if the participant develops symptoms during the delivery of the medication. The participant maybe admitted to the ward for further monitoring if symptoms become severe.

The effect of the study product on an unborn child is not known. The participants is advised to inform the study doctor immediately if she thinks that she is pregnant during the study. If she is pregnant, the study therapy will be discontinued immediately and she will be removed from the study. The participant is advised to ask the doctor if he/she needs more information on the risks and side effects. The trial staff will inform him/her in a timely manner about any new findings or changes about the study product which may affect his/her health or willingness to continue in this study. Where necessary, the participant may be asked to re-consent to participate.

All of the participant's information obtained in this study will be kept and handled in a confidential manner, in accordance with applicable laws and/or regulations. When publishing or presenting the study results, the participant's identity will not be revealed without his/her expressed consent. Individuals involved in this study, qualified monitors and auditors, the sponsor or its affiliates and governmental or regulatory authorities may inspect and copy his/her medical records, where appropriate and necessary. Data is kept in both hard and digital copies. Hard copies are kept in lockable cabinets with controlled access when not under direct supervision of a member of the research team. The study data is kept for at least 5 years and henceforth may be destroyed after the duration has expired.

The study doctor or the sponsor may due to concerns for the participant's safety, stop the study at any time. If the study is stopped early for any reason the participant will be informed and arrangements made for the participants future care.

Plan for data analysis and interpretation The raw data will be processed and entered for data analysis starting as soon as the patient is recruited till the end of the study.Data will be sorted out and processed on a weekly basis. Data entry, utilizing codes was done using SPSS software version 23. Computer assisted analysis will be carried out at the end of the study.

For the proposed study, sample size was determined by using power study. This power study was performed using web based sample size calculator (http://www.stat.ubc.ca/~rollin/stats/ssize/n2a.html) which is a very useful tool in medical and biological research to determine the sample size. Considering 90% power and 5% marginal error (type one error for α value=0.05), this study gives a minimum sample size of 55 per group (based on the mean and SD obtained from a recent study [13]). Finally, the investigators take 60 sample sizes per group.

Randomization was done by using a web based randomizer http://www.graphpad.com/quickcalcs/randomize1@ 18th March 2016@1500H where the total number is separated in 2 groups and each group containing 60 samples. The numbers are randomized and printed according to the web based randomizer at the aforementioned date and time. Generated numbers are then saved for further reference. The numbers are then placed in envelopes and given to the patient. The numbers which are received by the patient will determine the group by which the patient is selected into.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-40 years of age regardless of race of gender.
* Patients requiring the use of a rigid nasoendoscopy for the diagnosis of nasal pathology

Exclusion Criteria:

* Patients with underlying systemic medical problems. e.g. Bronchial Asthma, Chronic lung disease, Diabetes, Chronic Kidney disorder, Cerebrovascular accidents (CVA),SLE
* Patients who have nasal pathologies such as nasal polyps, inverted papillomas, malignancies, deviated nasal septums, septal perforations, deformed external nose, cleft palates.
* Patients with a history of nasal surgery
* Patients with a history of intranasal topical medications (E.g Intranasal oxymetazoline,)
* Patients who are pregnant and are breastfeeding.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Nasal resistance | Pre-procedure and 5,10,15 and 30 minutes after introduction of nasal spray/nebulizer
  Change in Nasal resistance in Pa/cm3/s

SECONDARY OUTCOMES:
Age | Pre-procedure
  Age in years
Gender | Pre-procedure
  Male/female
BMI | Pre-procedure
  Body Mass Index
VAS (Visual analogue score) pain score | Pre-procedure and 30 minutes after introduction of nasal spray/nebulizer
  VAS (Visual analogue score) pain score
nasal flow rate | Pre-procedure and 5,10,15 and 30 minutes after introduction of nasal spray/nebulizer
  nasal flow rate in ml/s

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - University of Malaya Medical center, Kuala Lumpur, Kuala Lumpur
  - Hospital Tengku Ampuan rahimah, Klang, Selangor

IPD SHARING:
Plan to Share IPD: No